CLINICAL TRIAL: NCT00599911
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, Active-referenced, Dose-finding Study of Lu AA24530 in Major Depressive Disorder
Brief Title: Dose-finding Study With Lu AA24530 in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11918A; 2007-001071-11 (EudraCT Number)
Record Dates: First submitted 2007-12-28; First posted 2008-01-24 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
Keywords: Drug therapy; Depressive disorder; Antidepressive agents; Depressive symptoms; Affective disorders; Randomized controlled trial; Placebo-controlled; Double-blind; Active reference; Multicenter study
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Mood Disorders | interventions — Tedatioxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lu AA24530: 5 mg (Experimental)
  Interventions: Drug: Lu AA24530
- Lu AA24530: 10 mg (Experimental)
  Interventions: Drug: Lu AA24530
- Lu AA24530: 20 mg (Experimental)
  Interventions: Drug: Lu AA24530
- Duloxetine: 60 mg (Active Comparator)
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AA24530 — per oral, once daily for 6 weeks
  Arms: Lu AA24530: 10 mg; Lu AA24530: 20 mg; Lu AA24530: 5 mg
Drug: Duloxetine — per oral, once daily for 6 weeks
  Arms: Duloxetine: 60 mg
Drug: Placebo — per oral, once daily for 6 weeks
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the efficacy in treating patients with Major Depressive Disorder of one or more doses of Lu AA24530 relative to placebo

DETAILED DESCRIPTION:
According to the World Health Organisation, Major Depressive Disorder is the leading cause of disability and the 4th leading contributor to the global burden of disease. There are unmet medical needs in the treatment of depressive disorders in terms of insufficient effectiveness and unpleasant side-effects of current therapies. The overall prognosis of the disorder is positive for the majority of patients, but as many as 30% of patients will develop a chronic and treatment-resistant depression. In the study, patients with depression are treated for 6 weeks. Assessments of efficacy and safety are taking place every week for the first 4 weeks and again after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Episode that has lasted at least 3 months
* Moderate to severe depression

Exclusion Criteria:

* Any current psychiatric disorder established as the principal diagnosis other than MDD as defined in the DSM-IV-TR and as assessed with the Mini-International Neuropsychiatric Interview (MINI)
* Current or past history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR
* Major Depressive Episode that has been unresponsive to two adequate courses of antidepressant treatment, each of at least 6 weeks duration
* Electroconvulsive therapy within 6 months prior to Baseline
* Ongoing formal cognitive or behavioural therapy, systematic psychotherapy, or plans to initiate such therapy during the study
* Clinically significant unstable illness, for example, hepatic or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic, or metabolic disturbance
* The patient is pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The difference in change from baseline to end of treatment on the Montgomery-Åsberg Depression Rating Scale total score | 6 weeks

SECONDARY OUTCOMES:
Response rate, remission rate, and safety | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (72):
- Australia (5):
  - AU002, Brisbane
  - AU001, Brisbane
  - AU003, Dandenc
  - AU004, Epping
  - AU006, Malvern
- Austria (3):
  - AT001, Vienna
  - AT002, Vienna
  - AT003, Vienna
- Belgium (2):
  - BE003, Diest
  - BE002, Sint-Niklaas
- Canada (5):
  - CA006, Mississauga
  - CA004, Oakville
  - CA003, Penticton
  - CA005, Toronto
  - CA001, Vancouver
- Czechia (6):
  - CZ002, Brno
  - CZ005, Prague
  - CZ001, Prague
  - CZ004, Prague
  - CZ003, Prague
  - CZ006, Sternberk
- Finland (6):
  - FI001, Helsinki
  - FI003, Helsinki
  - FI006, Jarvenpaa
  - FI004, Seinäjoki
  - FI005, Tampere
  - FI002, Turku
- France (7):
  - FR007, Angoulême
  - FR002, Dole
  - FR003, Montpellier
  - FR001, Orvault
  - FR008, Rouen
  - FR004, Savigny-sur-Orge
  - FR005, Wattigny
- India (6):
  - IN001, Ahmedabab
  - IN009, Ahmedabad
  - IN007, Chennai
  - IN006, Hyderabaad
  - IN003, Mangalore
  - IN002, Pune
- Lithuania (3):
  - LT002, Kaunas
  - LT003, Klaipėda
  - LT001, Vilnius
- Malaysia (2):
  - MY002, Kuala Lumpur
  - MY003, Kuala Lumpur
- Norway (3):
  - NO004, Fredrikstad
  - NO001, Hamar
  - NO003, Skien
- Philippines (3):
  - PH002, Las Piñas
  - PH003, Mandaluyong
  - PH001, Mandaue City
- Russia (5):
  - RU005, Arkhangelsk
  - RU002, Nikol'skoye
  - RU003, Saint Petersburg
  - RU004, Saratov
  - RU001, Tomsk
- Serbia (2):
  - RS004, Belgrade
  - RS002, Kragujevac
- South Korea (3):
  - KR003, Gwangju
  - KR002, Seoul
  - KR001, Seoul
- Sweden (6):
  - SE006, Halmstad
  - SE001, Linköping
  - SE002, Lund
  - SE003, Malmo
  - SE005, Stockholm
  - SE004, Uppsala
- Ukraine (5):
  - UA003, Dnipro
  - UA005, Kharkiv
  - UA002, Kyiv
  - UA004, Lviv
  - UA001, Odesa

REFERENCES:
- [Derived] Belzeaux R, Gorgievski V, Fiori LM, Lopez JP, Grenier J, Lin R, Nagy C, Ibrahim EC, Gascon E, Courtet P, Richard-Devantoy S, Berlim M, Chachamovich E, Theroux JF, Dumas S, Giros B, Rotzinger S, Soares CN, Foster JA, Mechawar N, Tall GG, Tzavara ET, Kennedy SH, Turecki G. GPR56/ADGRG1 is associated with response to antidepressant treatment. Nat Commun. 2020 Apr 2;11(1):1635. doi: 10.1038/s41467-020-15423-5. PMID 32242018
- [Derived] Belzeaux R, Fiori LM, Lopez JP, Boucekine M, Boyer L, Blier P, Farzan F, Frey BN, Giacobbe P, Lam RW, Leri F, MacQueen GM, Milev R, Muller DJ, Parikh SV, Rotzinger S, Soares CN, Uher R, Foster JA, Kennedy SH, Turecki G. Predicting Worsening Suicidal Ideation With Clinical Features and Peripheral Expression of Messenger RNA and MicroRNA During Antidepressant Treatment. J Clin Psychiatry. 2019 May 7;80(3):18m12556. doi: 10.4088/JCP.18m12556. PMID 31087825
- Available data/document: EMA EudraCT Results: 2007-001071-11 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2007-001071-11/results